CLINICAL TRIAL: NCT05020327
Title: Inpatient Penicillin Allergy Delabeling Pilot Project at University Hospitals-Rainbow Babies and Children's Hospital in Cleveland, Ohio
Brief Title: Inpatient Penicillin Allergy Delabeling Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Ankita Desai, Associate Professor, Director of Pediatric Antimicrobial Stewardship, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: STUDY20200136
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: Penicillin Allergy; Penicillin Sensitivity; Penicillin Reaction; Penicillin Intolerance
Keywords: Penicillin allergy; Penicillin delabeling
MeSH Terms: interventions — Electronic Health Records

STUDY DESIGN:
Intervention Model Description: Patients will be screened by questionnaire to determine No risk, Low risk, or High Risk for penicillin allergic reaction. Those that are deemed Low Risk based on questionnaire, will be subsequently challenged with graded oral amoxicillin challenge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Risk Patients (Experimental): This is the group of patients who will undergo the graded oral amoxicillin challenge testing. Total dose of the amoxicillin will be 45 mg/kg (maximum of 1000 mg). 10 % of this dose will be given first followed by 90 % of the dose 30 minutes after. Each dose will be given only once.
  Interventions: Drug: Graded Oral Amoxicillin Challenge; Other: De-labelling in electronic medical record; Other: Referral to Allergy Immunology/Retention of Allergy Label
- No Risk Patients (Other): Patients in the group will be de-labeled in the electronic medical record for No Risk for allergic reaction to amoxicillin based on screening questionnaire.
  Interventions: Other: De-labelling in electronic medical record
- High Risk (Other): Patients in this group are deemed high risk for allergic reaction to penicillin based on screening questionnaire and will remain labeled with allergy in the electronic medical record. They will be referred as outpatient to allergy-immunology for further evaluation.
  Interventions: Other: Referral to Allergy Immunology/Retention of Allergy Label

INTERVENTIONS:
Drug: Graded Oral Amoxicillin Challenge — Oral amoxicillin at 45 mg/kg (maximum of 1000 mg) to be divided into two doses: 10 % initial dose and then 90% remaining dose - doses will be separated by 30 minute interval
  Other Names: Amoxicillin Challenge
  Arms: Low Risk Patients
Other: De-labelling in electronic medical record — Patients with No Risk for allergic reaction will be de-labelled for allergy in the electronic medical record.
  Arms: Low Risk Patients; No Risk Patients
Other: Referral to Allergy Immunology/Retention of Allergy Label — Patients deemed to be High Risk for allergic reaction will be referred to Allergy Immunology as outpatient and allergy label will be retained.
  Arms: High Risk; Low Risk Patients

SUMMARY:
The study will identify pediatric patients 3-18 years old who have penicillin allergy label in the electronic medical record. Those who are identified will be stratified into no-risk, low-risk and high-risk category using a screening questionnaire. The following definitions will be followed:

No-risk: Patients who are historically labeled with penicillin allergy in the EMR based on family history alone OR those who have tolerated penicillin after a concerning incident without any reaction OR with penicillin allergy label but deny any history of reaction to any form of penicillin on screening questionnaire

Low-risk: Patients with previous reaction not suggestive of anaphylaxis (defined below) AND not requiring hospitalization for the reaction OR reaction considered non- immunologic (e.g. diarrhea, nausea, yeast vaginitis) OR exposure to penicillin- containing antibiotic after the date of reported reaction with no anaphylaxis and hospitalization AND no serious types of delayed reactions such as Steven- Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), acute interstitial nephritis (AIN), drug-induced hepatitis or other documented organ injury, drug rash eosinophilia systemic symptoms (DRESS), hemolytic anemia, drug-induced cytopenia, and serum sickness. Patients who had delayed reaction (onset more than 24 hours) of isolated, non-progressive symptoms (such as rash/hives alone) also belong to this group.

High-risk: Patients with penicillin allergy label on EMR with previous reaction suggestive of anaphylaxis (defined below) OR requiring hospitalization/epinephrine administration for the reaction OR reactions considered immunologic (angioedema, joint pains) OR involving serious types of reactions such as Steven-Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), acute interstitial nephritis (AIN), drug-induced hepatitis or other documented organ injury, drug rash eosinophilia systemic symptoms (DRESS), hemolytic anemia, drug-induced cytopenia, and serum sickness. Patients who were previously diagnosed with penicillin allergy by an allergist also belong to the high-risk group.

Patients in the no-risk group will be immediately delabeled. Patients in the high-risk group will be referred to allergy/immunology for further work up. The focus of this study is to identify the patients who belong to the low-risk group. This group of patients will be subjected to graded oral amoxicillin challenge testing. Those who will have reactions compatible with allergy will have their allergy status retained in the electronic medical record. Those that will not have reactions or those that will have reactions that are not compatible with allergy will be delabeled in the electronic medical record.

DETAILED DESCRIPTION:
A. Specific Aims and Hypotheses

General Objective:

To verify pediatric patients with reported penicillin allergy in electronic medical record (EMR) by performing direct oral amoxicillin challenge testing.

Hypothesis: Pediatric patients with reported penicillin allergy in EMR can be verified by performing direct oral amoxicillin challenge testing.

Specific objectives:

1. To identify no-risk, low-risk and high-risk patients among pediatric patients with reported penicillin allergy in EMR through a questionnaire.

   Hypothesis: No-risk, low-risk and high-risk pediatric patients with reported penicillin allergy in EMR can be identified using a questionnaire.
2. To be able to delabel pediatric patients with reported penicillin allergy in EMR who are identified as no-risk.

   Hypothesis: No-risk pediatric patients with reported penicillin allergy in EMR can be delabeled using a questionnaire.
3. To be able to delabel identified low-risk pediatric patients with reported penicillin allergy in EMR who are verified not allergic to penicillin by direct oral amoxicillin challenge testing.

   Hypothesis: Identified low-risk pediatric patients with reported penicillin allergy in EMR using a questionnaire can be verified using direct oral amoxicillin challenge testing.
4. To be able to provide proper referral guidance to patients identified as high-risk and those who failed oral amoxicillin challenge testing to allergy and immunology for further evaluation and management.

Hypothesis: Proper referral guidance to patients identified as high-risk and those who failed oral penicillin challenge testing to allergy and immunology can be provided for their further evaluation and management.

B. Background and Significance Penicillin remains a reliable class of antibiotics that addresses a majority of infections both in outpatient and inpatient settings.(1,2) It is also one of the cheapest antibiotics to use for empiric therapy for susceptible infections.(3,4) Emerging literature suggests that the number of patients with historical penicillin allergy is an overestimate. A growing number of studies show that only approximately 1-10 % of patients with historical penicillin allergy are truly allergic after verified allergy testing is done.(1-3,5,7,8,10,11,12) Despite this, efforts on antibiotic allergy delabeling remains sparse and penicillin allergy remains to be the most common drug allergy reported.

Few institutions have implemented, much less conceptualized, protocols to determine truly allergic patients who have reported penicillin allergy when diagnosed with infections theoretically susceptible to penicillin.(6) One limitation perhaps is the absence of validated questionnaire that uniformly captures accepted levels of risk especially in the pediatric population.(7) As a result, these patients end up receiving alternative antimicrobial agents that pose a risk for emergence of resistance, development of unnecessary intestinal dysbiosis, and increased economic burden to health care resulting in suboptimal clinical outcome. (1-6) Studies aiming to validate direct oral challenge testing as a means of penicillin allergy delabeling is a fertile avenue for this clinical query to be addressed in a cost-effective and timely manner. (8-13)

Identifying patients with no immunologically-mediated penicillin allergy and delabeling them in the electronic medical record (EMR) accordingly will mitigate the use of second-line antibiotics, aid in minimizing development of antimicrobial resistance, ameliorate unnecessary economic burden, and overall lead to positive impact in clinical outcome and patient care. (1,5,7,8,10,11,12) In the same way, this process will also identify patients with true penicillin allergy creating a point-of-care opportunity to provide them proper guidance on the importance of Allergy/Immunology follow-up for further evaluation and management.

C. Methods

Population of Interest:

Patients 3-18 years old admitted at our institution will be screened for inclusion. We will screen approximately 800 patients and enroll 60 patients in our study (based on the weekly census) over a span of 3 months. HIPAA regulations will be strictly observed in data handling to protect patient privacy.

Screening and consenting of patients:

Signed parental consent and verbal consent from study team will be obtained prior to screening. Patients will be screened using a questionnaire to identify risk status. Patients identified as no-risk (EMR label based purely on family history of penicillin allergy, mislabeled patients) will be immediately delabeled in EMR. High-risk patients (those with reaction consistent with IgE mediated reaction or with history of anaphylaxis) will be excluded. Guidance on further care such as referral to an allergist will be recommended if not yet done. Low-risk patients (those with mild reaction not consistent with IgE mediated reaction, no history of serious delayed reaction or no reaction on subsequent penicillin receipt) will be identified to undergo graded direct oral amoxicillin challenge testing.

Oral Amoxicillin Challenge Testing:

Signed parental consent and patient assent (7 years and older) will be obtained prior to challenge testing. Only low-risk patients with parent/guardian in the room and no receipt of anti-histamine 48 hours prior will be challenged. Only patients who can tolerate enteral amoxicillin will be challenged. Rescue kits (containing diphenhydramine, epinephrine and albuterol) will be ready at bedside prior to challenging. Baseline vital signs will be obtained prior to challenging. Oral challenge testing will be graded: initial 10% of the dose followed by remaining 90% of the dose (total dose 45 mg/kg with maximum of 1000 mg) 30 minutes apart. Vital signs will be repeated 30 minutes after the first dose, 30 minutes after the second dose and finally 60 minutes after the second dose. Study team will administer amoxicillin doses and monitor for signs of amoxicillin allergic reaction. Any reaction during the testing will be assessed by trained study team member. A clinical event note will be written in the EMR for any reaction occurring during the testing as well the management implored to mitigate reaction.

Delabeling:

Low-risk patients who passed the challenge testing will be delabeled in EMR. Documentation of the result will be sent to patient's primary care doctor (with permission from parent) for guidance on future use of penicillin.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for screening

* Patients 3-18 years old admitted at our institution with penicillin allergy label in electronic medical record
* Patients with available parent/s or legal guardian who can give both written and verbal consent to the oral challenge testing
* Patients with available parent/s or legal guardian during the conduct of oral amoxicillin challenge testing

Inclusion Criteria for oral challenge test

- Patients who will be identified as low-risk patients based on the standardized screening questionnaire. Low-risk group patients are those patients with previous reaction not suggestive of anaphylaxis AND not requiring hospitalization for the reaction OR reaction considered non-immunologic (e.g. diarrhea, nausea, yeast vaginitis) OR exposure to penicillin-containing antibiotic after the date of reported reaction with no anaphylaxis and hospitalization AND no serious types of delayed reactions such as Steven-Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), acute interstitial nephritis (AIN), drug-induced hepatitis or other documented organ injury, drug rash eosinophilia systemic symptoms (DRESS), hemolytic anemia, drug-induced cytopenia, and serum sickness. - ---- Patients who had delayed reaction (onset more than 24 hours) of isolated, non-progressive symptoms (such as rash/hives alone) also belong to this group.

Exclusion Criteria:

Exclusion Criteria for screening

* Patients who cannot tolerate amoxicillin/penicillin by enteral route.
* Patients with no parents or legal guardian available to give both written and verbal consent to the oral challenge testing
* Patients with no available parents or legal guardian during the conduct of oral amoxicillin challenge testing
* Patients currently on antihistamine or have received antihistamine in the previous 48 hours
* Patients who are critically ill
* Patients who have been vomiting more than twice in the past 24 hours or are actively vomiting
* Patients with respiratory symptoms warranting oxygen therapy or pulmonary finding of wheezing or stridor
* Patients identified as having anaphylactic reaction to penicillin in the electronic medical record

Exclusion Criteria for oral challenge testing

* Patients who will be identified as no-risk patients based on the standardized screening questionnaire. No-risk group patients are those patients who are historically labeled with penicillin allergy in the EMR based on family history alone OR those who have tolerated penicillin after a concerning incident without any reaction OR with penicillin allergy label but deny any history of reaction to any form of penicillin on screening questionnaire
* Patients who will be identified as high-risk patients based on the standardized screening questionnaire. High-risk group patients are those patients with penicillin allergy label on EMR with previous reaction suggestive of anaphylaxis OR requiring hospitalization/epinephrine administration for the reaction OR reactions considered immunologic (angioedema, joint pains) OR involving serious types of reactions such as Steven-Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), acute interstitial nephritis (AIN), drug-induced hepatitis or other documented organ injury, drug rash eosinophilia systemic symptoms (DRESS), hemolytic anemia, drug-induced cytopenia, and serum sickness. Patients who were previously diagnosed with penicillin allergy by an allergist also belong to the high-risk group.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ankita Desai, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vyles D, Adams J, Chiu A, Simpson P, Nimmer M, Brousseau DC. Allergy Testing in Children With Low-Risk Penicillin Allergy Symptoms. Pediatrics. 2017 Aug;140(2):e20170471. doi: 10.1542/peds.2017-0471. Epub 2017 Jul 3. PMID 28674112
- [Result] du Plessis T, Walls G, Jordan A, Holland DJ. Implementation of a pharmacist-led penicillin allergy de-labelling service in a public hospital. J Antimicrob Chemother. 2019 May 1;74(5):1438-1446. doi: 10.1093/jac/dky575. PMID 30753497
- [Result] Blumenthal KG, Ryan EE, Li Y, Lee H, Kuhlen JL, Shenoy ES. The Impact of a Reported Penicillin Allergy on Surgical Site Infection Risk. Clin Infect Dis. 2018 Jan 18;66(3):329-336. doi: 10.1093/cid/cix794. PMID 29361015
- [Result] Au LYC, Siu AM, Yamamoto LG. Cost and Risk Analysis of Lifelong Penicillin Allergy. Clin Pediatr (Phila). 2019 Oct;58(11-12):1309-1314. doi: 10.1177/0009922819853014. Epub 2019 Jun 19. PMID 31216862
- [Result] Sagar PS, Katelaris CH. Utility of penicillin allergy testing in patients presenting with a history of penicillin allergy. Asia Pac Allergy. 2013 Apr;3(2):115-9. doi: 10.5415/apallergy.2013.3.2.115. Epub 2013 Apr 26. PMID 23667835
- [Result] Arnold A, Sommerfield A, Ramgolam A, Rueter K, Muthusamy S, Noble V, von Ungern-Sternberg BS, Lucas M. The role of skin testing and extended antibiotic courses in assessment of children with penicillin allergy: An Australian experience. J Paediatr Child Health. 2019 Apr;55(4):428-432. doi: 10.1111/jpc.14220. Epub 2018 Sep 13. PMID 30209846
- [Result] Shenoy ES, Macy E, Rowe T, Blumenthal KG. Evaluation and Management of Penicillin Allergy: A Review. JAMA. 2019 Jan 15;321(2):188-199. doi: 10.1001/jama.2018.19283. PMID 30644987
- [Result] Kuruvilla M, Shih J, Patel K, Scanlon N. Direct oral amoxicillin challenge without preliminary skin testing in adult patients with allergy and at low risk with reported penicillin allergy. Allergy Asthma Proc. 2019 Jan 1;40(1):57-61. doi: 10.2500/aap.2019.40.4184. PMID 30582497
- [Result] Graham F, Tsabouri S, Caubet JC. Hypersensitivity reactions to beta-lactams in children. Curr Opin Allergy Clin Immunol. 2018 Aug;18(4):284-290. doi: 10.1097/ACI.0000000000000453. PMID 29870460
- [Result] Mustafa SS, Conn K, Ramsey A. Comparing Direct Challenge to Penicillin Skin Testing for the Outpatient Evaluation of Penicillin Allergy: A Randomized Controlled Trial. J Allergy Clin Immunol Pract. 2019 Sep-Oct;7(7):2163-2170. doi: 10.1016/j.jaip.2019.05.037. Epub 2019 Jun 4. PMID 31170542
- [Result] Moral L, Caubet JC. Oral challenge without skin tests in children with non-severe beta-lactam hypersensitivity: Time to change the paradigm? Pediatr Allergy Immunol. 2017 Dec;28(8):724-727. doi: 10.1111/pai.12800. Epub 2017 Oct 3. PMID 28892222
- [Result] Kelso JM. Provocation Challenges to Evaluate Amoxicillin Allergy in Children. JAMA Pediatr. 2016 Jun 6;170(6):e160282. doi: 10.1001/jamapediatrics.2016.0282. Epub 2016 Jun 6. No abstract available. PMID 27043299
- [Result] Mill C, Primeau MN, Medoff E, Lejtenyi C, O'Keefe A, Netchiporouk E, Dery A, Ben-Shoshan M. Assessing the Diagnostic Properties of a Graded Oral Provocation Challenge for the Diagnosis of Immediate and Nonimmediate Reactions to Amoxicillin in Children. JAMA Pediatr. 2016 Jun 6;170(6):e160033. doi: 10.1001/jamapediatrics.2016.0033. Epub 2016 Jun 6. PMID 27043788
- [Result] Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol. 2006 Feb;117(2):391-7. doi: 10.1016/j.jaci.2005.12.1303. PMID 16461139
- [Result] Lieberman P, Nicklas RA, Randolph C, Oppenheimer J, Bernstein D, Bernstein J, Ellis A, Golden DB, Greenberger P, Kemp S, Khan D, Ledford D, Lieberman J, Metcalfe D, Nowak-Wegrzyn A, Sicherer S, Wallace D, Blessing-Moore J, Lang D, Portnoy JM, Schuller D, Spector S, Tilles SA. Anaphylaxis--a practice parameter update 2015. Ann Allergy Asthma Immunol. 2015 Nov;115(5):341-84. doi: 10.1016/j.anai.2015.07.019. No abstract available. PMID 26505932
- [Result] Bauer ME, MacBrayne C, Stein A, Searns J, Hicks A, Sarin T, Lin T, Duffey H, Rannie M, Wickstrom K, Yang C, Bajaj L, Carel K. A Multidisciplinary Quality Improvement Initiative to Facilitate Penicillin Allergy Delabeling Among Hospitalized Pediatric Patients. Hosp Pediatr. 2021 May;11(5):427-434. doi: 10.1542/hpeds.2020-001636. Epub 2021 Apr 13. PMID 33849960

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Risk Patients | No Risk Patients | High Risk
Started | 28 | 6 | 6
Completed | 12 | 5 | 6
Not Completed | 16 | 1 | 0
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — personal/cultural, ineligible | 12 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk Patients | No Risk Patients | High Risk | Total
Number analyzed (Participants) | 28 | 6 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.64 (4.44) | 13 (4.9) | 12.17 (4.383) | 11.23 (4.538)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 1 | 17
  Male | 15 | 3 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 28 | 6 | 6 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 28 | 6 | 6 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Allergy Status
Description: Participants with penicillin allergy status verification based on questionnaire and challenge
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk Patients | No Risk Patients | High Risk
Number analyzed (Participants) | 28 | 6 | 6
Participants | 28 | 6 | 6

2. Secondary Outcome: Number of Participants With no Penicillin Allergy Confirmed and De-labelled of Penicillin Allergy Based on Results of Questionnaire.
Description: Identification and delabeling of patients with no-risk status. These are the patients with no grounded history of reaction compatible with allergic reaction.
Time Frame: 3 hours
Population: Participants were not de-labeled after the questionnaire if they did not want to be de-labeled
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk Patients | No Risk Patients | High Risk
Number analyzed (Participants) | 28 | 6 | 6
Participants | 11 | 5 | 0

3. Secondary Outcome: Number of Participants Categorized as Low Risk for Penicillin Allergy Reaction With Confirmed True Penicillin Allergy as Measured by Failed Oral Amoxicillin Challenge
Description: Identification of patients who are low-risk with verified true allergy triggering referral to allergy immunology
Time Frame: 3 hours
Population: Data was not collected/analyzed for the "No Risk Patients" or "High Risk".
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk Patients | No Risk Patients | High Risk
Number analyzed (Participants) | 28 | 0 | 0
Participants | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With Confirmed True Allergy Without Challenge
Description: Identification of patients who are high risk. These are patients identified with history of reactions compatible with true allergy. Those who are not following with allergy can be given proper referral for further evaluation and management.
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk Patients | No Risk Patients | High Risk
Number analyzed (Participants) | 28 | 6 | 6
Participants | 0 | 0 | 6

ADVERSE EVENTS:
Time Frame: 6 months
Description: Reaction during oral challenge
Arm/Group | Low Risk Patients | No Risk Patients | High Risk
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/28 | 0/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Risk Patients (N=28) | No Risk Patients (N=6) | High Risk (N=6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT05020327/Prot_SAP_001.pdf